CLINICAL TRIAL: NCT05622617
Title: Prospective Observational Investigation of Serum Interleukin-20 Level and Paclitaxel-Associated Neuropathy in Breast Cancer Patients Receiving Paclitaxel Chemotherapy
Brief Title: Relationship Between Serum Interleukin-20 Level and Paclitaxel-associated Neuropathy
Acronym: NEUROTOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, Asoc Prof., Namik Kemal University
Other Study IDs: NEUROTOX
Record Dates: First submitted 2022-10-02; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Neuropathy Associated With Dysproteinaemias
Keywords: paclitaxel; peripheral neuropathy; Peripheral Neuropathy Induced by Paclitaxel
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: no intervention — no intervention

SUMMARY:
This study aims to investigate the correlation between paclitaxel-induced neuropathy and the measurement values of serum IL-20 levels at baseline and during chemotherapy in patients who will receive neoadjuvant or adjuvant paclitaxel chemotherapy with the diagnosis of early-stage or locally advanced breast cancer

DETAILED DESCRIPTION:
* Patients with the diagnosis of breast cancer who will be started on adjuvant or neoadjuvant paclitaxel chemotherapy will be included in the study.
* Patients who will receive standard breast cancer treatment (4 cycles of cyclophosphamide 600mg/m2 every 21 days + epirubicin 90mg/m2 followed by weekly paclitaxel 80 mg/m2 x 12 sessions) will be included in the study.
* Age, gender, additional disease, diagnosis dates, previous diseases and breast cancer subtypes of the patients who signed the informed consent form will be obtained from the electronic information system or by asking face-to-face.
* Serum IL-20 level will be studied from blood tests taken for routine chemotherapy. no extra blood sample will be taken for the study
* Neuropathy assessment will be evaluated with Organisation for Research and Treatment of Cancer (EORTC) chemotherapy-induced peripheral neuropathy (QLQ-CIPN20) Questionnaire, the sensitivity, and specificity of which have previously been demonstrated for chemotherapy-induced neuropathy. The Turkish validation questionnaire of the study, which was made before, will be conducted by the physician in charge before the paclitaxel chemotherapy and at the 1st and 12th weeks after the treatment, by asking the patient face to face.
* patients with diabetes mellitus and patients who had a history of peripheral neuropathy will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving paclitaxel chemotherapy for local advanced or early-stage breast cancer
* >18 years

Exclusion Criteria:

* advanced stage breast cancer
* having before peripheral neuropathy
* patients with diabetes mellitus
* < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only the female gender will be enrolled
Study Population: Patients receiving standard breast cancer treatment containing taxane
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Relationship with paclitaxel associated neuropathy and serum IL-20 level | January 01,2022 -December 31, 2022 is the deadline for patient inclusion
  Neuropathy measurement will be made face-to-face by the attending physician with a European Organisation for Research and Treatment of Cancer (EORTC) Chemotherapy-induced peripheral neuropathy (CIPN) Questionnaire after the first week after paclitaxel chemotherapy and the last week of 12 cycles of treatment
Relationship with paclitaxel associated neuropathy and serum IL-20 level | December 31, 2022 is the deadline for patient inclusion
  Neuropathy measurement will be made face-to-face by the attending physician with a European Organisation for Research and Treatment of Cancer (EORTC) Chemotherapy-induced peripheral neuropathy (CIPN) Questionnaire after the first week after paclitaxel chemotherapy and the last week of 12 cycles of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdag Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No